CLINICAL TRIAL: NCT05593796
Title: The Efficacy of Cognitive Behavioral Therapy(CBT) in Treatment of Methamphetamine Use Disorder
Brief Title: Cognitive Behavioral Therapy(CBT) in Treatment of Methamphetamine Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Tharwat Ahmad, Assistant lecture, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 715715
Record Dates: First submitted 2022-10-24; First posted 2022-10-25 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Methamphetamine Abuse
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: In phase 0:
  . These patients will undergo toxicological and psychiatric assessment and will be screened using the inclusion and exclusion criteria.
  phase 1:
  treatment-as-usual (TAU)- Group offered usual treatment include detoxification, medical care. Clinician-delivered CBT-Group offered 12 weekly, individual sessions of manual-guided CBT (15) delivered by trained clinician .
  phase2: a follow-up at 3-month post treatment phase without treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment-as-usual (TAU) (Active Comparator)
  Interventions: Behavioral: cognitive behavioral therapy
- Clinician-delivered CBT with tratment as usual (Active Comparator)
  Interventions: Behavioral: cognitive behavioral therapy

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — 12 weekly, individual sessions of manual-guided CBT delivered by trained clinician .

SUMMARY:
The efficacy of cognitive behavioral therapy(CBT) in treatment of methamphetamine use disorder

DETAILED DESCRIPTION:
Methamphetamine (MA) use is a serious public health concern in many countries and is second to cannabis as the most widely abused illicit drug in the world.

Over the past few years; there is an alarming increase in crystal methamphetamine (Shabu) abuse in the Egyptian market and The Egyptian government is annoyed from this issue because youth within the age of productivity were targeted.

Regular methamphetamine use can be associated with a range of psychiatric symptoms, particularly psychosis, anxiety, and depression.

No FDA approved pharmacological treatments are available for Meth addiction up till now and despite great advances achieved in understanding the neurobiology of drug addiction, the therapeutic options are severely limited . Consequently, the only available treatment at present is psychosocial intervention.

The effectiveness of CBT for other substance-use disorders (e.g. alcohol-, opioid- and cocaine-use disorders) has been well documented and as such this basic treatment approach has been applied to amphetamine-type stimulant (ATS)-use disorder .

Currently, there is not enough evidence to establish the efficacy of CBT for amphetamine -type stimulant( ATS) -use disorders because of a paucity of high-quality research in this area.

The present study will examine the efficacy of Cognitive behavioral therapy in reducing methamphetamine use in comparison to medical treatment usually taken in methamphetamine use disorder

ELIGIBILITY:
Inclusion Criteria:

* patients who meet the criteria for methamphetamine use disorder according to Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM 5) (10)
* aged of 15-49 years' old
* more than 9 year of education
* urine drug screening positive for methamphetamine

Exclusion Criteria:

* other Axis I disorder of DSM-V criteria such as bipolar disorder, schizophrenia, depression
* Had a legal case pending resulting in inability to commit to 12 weeks of treatment.
* Refusal to participate
* poly drug dependence.

Ages: 15 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
increase in the addiction severity index for methamphetamine use disorder | 12 weeks
  0-1 No imminent problem 2-3 slight problem 4-5 moderate problem 6-7considerable difficulty

IPD SHARING:
Plan to Share IPD: Undecided